CLINICAL TRIAL: NCT00002484
Title: A PHASE I TRIAL OF DOSE ESCALATION OF EXTERNAL BEAM RADIATION THERAPY USING CONFORMAL 3-DIMENSIONAL TREATMENT PLANNING FOR NON-SMALL CELL LUNG CANCER
Brief Title: Radiation Therapy Using 3-Dimensional Treatment Planning in Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91-121; CDR0000077300 (Registry Identifier: PDQ (Physician Data Query)); NCI-V91-0198
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

ARMS (1):
- external beam radiotherapy (Experimental): Patients undergo 3-dimensional conformal external beam radiotherapy 5 days a week for 8-10 weeks.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Computer systems that allow doctors to create a 3-dimensional picture of the tumor in order to plan treatment may result in more effective radiation therapy.

PURPOSE: Phase I trial to study the effectiveness of high-dose radiation therapy planned using a 3-dimensional picture of the tumor in treating patients who have stage I, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum dose of external beam irradiation deliverable using conformal 3-dimensional treatment planning in patients with non-small cell lung cancer.
* Determine the feasibility and efficacy of 3-dimensional treatment planning in delivering high doses of external beam radiotherapy to these patients.
* Determine whether computer-generated dose-volume histograms and normal tissue complication probability models can predict the degree of pulmonary toxicity resulting from external beam radiotherapy.
* Determine the relationship between dose of external beam radiotherapy and the degree of pulmonary function change.

OUTLINE: This is a dose escalation study.

Patients undergo 3-dimensional conformal external beam radiotherapy 5 days a week for 8-10 weeks.

Cohorts of 10 patients receive escalating doses of radiotherapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 20% of patients experience dose-limiting toxicity.

Patients are followed at 1 month and then every 4 months thereafter.

PROJECTED ACCRUAL: A total of 60-70 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Clinical stage T1-4, N0-2, M0

    * Clinical stage T1-2, N0-1 must be medically inoperable
* No distant metastases on history and physical exam, CBC, screening profile, CT or MRI of brain, CT of chest and abdomen (including adrenals and liver), and bone scan
* No pleural effusions
* Atelectasis not clearly distinguishable from tumor mass allowed provided all tumor and atelectasis together represent a volume that can be safely treated to the total dose delivered to gross disease
* Diffuse pulmonary infiltrates thought to represent benign disease allowed only if representative lesion samples are proven by biopsy or cytology not to contain cancer
* No diffuse bronchoalveolar carcinoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other malignancy within the past 5 years except nonmelanomatous skin cancer or noninvasive cervical carcinoma
* No other medical illness that cannot be adequately controlled with appropriate therapy or that is considered severe enough to preclude a radical treatment approach

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for lung cancer

Chemotherapy

* No prior chemotherapy for lung cancer

Endocrine therapy

* No prior endocrine therapy for lung cancer

Radiotherapy

* No prior radiotherapy for lung cancer

Surgery

* No prior surgery for lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 1991-10; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Determine the maximum dose of external beam irradiation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Rosenzweig, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Armstrong J, Raben A, Zelefsky M, Burt M, Leibel S, Burman C, Kutcher G, Harrison L, Hahn C, Ginsberg R, Rusch V, Kris M, Fuks Z. Promising survival with three-dimensional conformal radiation therapy for non-small cell lung cancer. Radiother Oncol. 1997 Jul;44(1):17-22. doi: 10.1016/s0167-8140(97)01907-5. PMID 9288852
- [Result] Armstrong J, Zelefsky M, Burt M, et al.: Acute toxicity of high dose 3-dimensional conformal radiation therapy (3-DCRT) for non small-cell lung cancer (NSCLC). [Abstract] Proceedings of the American Society of Clinical Oncology 12: A-1171, 348, 1993.